CLINICAL TRIAL: NCT04877704
Title: The Effect of Symprove, a Multi-strain Probiotic, as an Adjuvant in the Management of COVID-19 in Hospitalized Patients
Brief Title: Symprove (Probiotic) as an add-on to COVID-19 Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 290407
Record Dates: First submitted 2021-05-05; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symprove (Experimental): Symprove probiotic
  Interventions: Other: Symprove (probiotic)
- Placebo (Placebo Comparator): Matched placebo provided by Symprove. Identical in appearance to Symprove probiotic.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Symprove (probiotic) — Symprove's unique water-based formula is packed full of live, active bacteria. It is a probiotic, not a drug.
  Arms: Symprove
Other: Placebo — Matched placebo to Symprove probiotic
  Arms: Placebo

SUMMARY:
The major impact of COVID-19 has been that the severity of respiratory symptoms require intensive hospital treatment. There is significant mortality and many of the survivors have a delayed recovery requiring intensive prolonged rehabilitation.

COVID-19 is a multi-systemic disease in which different mechanisms within the body are affected; including the 'Gut microbiome'. 'Gut microbiome' refers to the bacteria living in intestines. While some bacteria is harmful, many are extremely beneficial and necessary for a healthy body. Many patients have gastrointestinal symptoms and there is a major change in the gut micro flora (microbiome), which may have an adverse effect on the respiratory symptoms. The probiotic, Sivomix, was given to hospitalized COVID-19 patients was associated with a more rapid recovery in gastrointestinal symptoms on day 3 and 7, and an eight fold reduction in the requirement for mechanical ventilation in an open trial.

This is a randomized clinical trial, with a recruitment target of 60 patients admitted with COVID-19 symptoms to the general medical wards. Patients will be randomized to receive the probiotic, Symprove, or placebo in addition to their standard of care treatment. Patients will need take either probiotic/placebo daily for 3 months. All follow-up will be whilst they are an inpatient or as a telephone follow-up; they will not need to attend at the hospital to participate.

There is a biological sub-study incorporated into the protocol, but participation is optional. If patients consent to this, they will also need to provide blood, faecal and saliva samples at baseline, Day 7 and final visit (3 months after randomisation). Patients who consent to providing biological samples will need to visit the hospital at Day 7 and final visit.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients who are hospitalised with respiratory COVID-19
* Ability to give informed consent
* Aged 20-85

Exclusion Criteria:

* Patients not meeting the inclusion criteria that have COVID-19
* Inability to consent
* Pregnancy
* Severe pre-existing mental health disorders or addictions

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-31 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | 12 months
  To assess if taking the probiotic Symprove reduces the length of hospital stay of patients with symptomatic respiratory COVID-19 infection

SECONDARY OUTCOMES:
Clinical symptoms | 7 days
  Whether administration of Symprove is associated with significantly greater improvements in clinical symptoms as opposed to placebo on day 3 and 7.
Intestinal inflammation | 3 months
  Whether Symprove reduced intestinal inflammation as compared with that seen in placebo are improved (at day 7 and 3 months).
Symptom recovery | 3 months
  Whether symptom recovery is more complete with the probiotic 3 months from the onset of the trial (all subjects will receive Symprove or placebo for 3 months).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver Studies, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No